CLINICAL TRIAL: NCT03081637
Title: Filamin A Expression in HCC Patients
Brief Title: FLNA in HCC Patients
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Professor of Surgery, Director Department of Hepatobiliary and General Surgery, University of Milan
Other Study IDs: FLNA in HCC
Record Dates: First submitted 2017-03-02; First posted 2017-03-16 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Surgical specimen from patients resected for HCC.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The risk of recurrence after hepatectomy for hepatocellular carcinoma (HCC) is very high. Having a predictive marker of early recurrence (ER) would be desirable to personalize the follow-up and possibly develop new targeted therapy. The aim of this study was to test the expression of Filamin A (FLNA) in a cohort of patients operated for HCC.

DETAILED DESCRIPTION:
A consecutive cohort of resected HCC patients will be analyzed. Several different prognostic factors, including FLNA expression, will be tested against the risk of ER. FLNA expression will be analyzed with immunohistochemistry in the intra-tumoral and extra-tumoral tissue compartments using a dedicated tissue microarray.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were represented by the histological positivity for HCC with complete clinical, surgical, pathological, and follow-up data.

Exclusion Criteria:

* Patients preoperatively treated with chemotherapy or trans-arterial therapy were excluded.
* Similarly, patients operated for recurrent HCC or with non-radical surgery or with missing data were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients submitted to hepatectomy at our unit in the above mentioned frame time.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Rate of expression of Filamin A (FLNA) in HCC specimens from patients resected for HCC. | 2 years after surgery as a minimum follow-up
  The rate of expression of FLNA in HCC specimens will be measured using standard immunohistochemistry methodology on surgical specimens. Such expression rate will be correlated to several different clinical and pathological parameters.